CLINICAL TRIAL: NCT00812864
Title: Pharmacokinetic Study of Capecitabine in Elderly Cancer Patient (≥75 Years)
Brief Title: Pharmacokinetic Study of Capecitabine in Elderly Cancer Patient (≥ 75 Years)
Acronym: capagec
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I07028; N° EudraCT : 2008-001195-7
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2009-09

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Capecitabine; pharmacocinetics; Breast metastatic cancer; colorectal metastatic cancer; Elderly patients
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine (Experimental)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Pharmacokinetic of its metabolites.
  Capecitabine, 1250 mg/m2 twice a day

SUMMARY:
The aim of the study is to determine blood concentration evolution of capecitabine and its active metabolites, in elderly patient 75 years and more.

DETAILED DESCRIPTION:
Blood samples will be taken before 1rst course of chemotherapy of capécitabine for colorectal or breast metastatic cancer.

Pharmacokinetic will be realizes at several times (H0,5, H1, H1,5, H2, H4, H6, H8) and repeated at D14 of the 2d cycle

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients 75 years old or more
* Life expectancy of greater then or equal to 6 months
* Histologically proven metastatic breast or colorectal cancer, requiring a chemotherapy by capecitabine according to the habitual schema
* Metastatic situation whatever treatment line
* Previous hormonotherapy for breast cancer, prior chemotherapy (without capecitabine) in adjuvant and/or metastatic indication (colorectal or breast cancer), or radiotherapy (colorectal or breast cancer) are allowed
* One or more measurable target lesion (RECIST criteria)
* ADL>4 (geriatric scales)
* GSD<12 (geriatric scales)
* Laboratory values :
* creatinine clearance (CrCl) >=30 mL/min according to Cockcroft formula
* Adequate bone marrow function (neutrophils count > 1.5 x 10^9/L, platelets > 100 x 10^9/L, hemoglobin [Hb] > 10g/dl)
* Adequate hepatic function: total bilirubin < 1,5 x upper normal limit, aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) < 2,5x upper normal limits (in case of liver metastases < 5 x upper normal limits)
* Alcalin phosphatases <=2,5x ULN (<=5 x ULN if liver metastases present).
* Subjects must be willing to be followed during the course of treatment/observation and follow-up.
* Signed written informed consent before first course of chemotheray

Exclusion Criteria:

* Age < 75 years
* known brain metastases
* Concomitant oncologic treatment ongoing
* History of severe or unscheduled reaction to fluoropyrimidine treatment
* Prior unanticipated severe reaction to capecitabine or metabolites and to fluoropyrimidine therapy
* Patient with leucopenia
* sorivudine or chemical analogues treatment like brivudine
* Physiological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Concomitant severe affections wich lead life expectancy inferior to 3 monthes
* Uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure, coronarian spasmes
* No possible oral administration
* known DPD deficiency
* Treatment with experimental therapy ongoing or within four weeks before inclusion.
* Other cancers within the last five years, with the exception of adequately treated cone-biopsied in situ carcinoma of the uterin cervix or basal or squamous cell carcinoma of the skin

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Mean value and dispersion of the main plasmatics pharmacokinetics parameters of capécitabine, 5'DFUR, 5-FU and FBAL. | 1 year
  pharmacokinetics of capécitabine

SECONDARY OUTCOMES:
Adverse effects evaluation after every course of chemotherapy according to NCI criteria during 6 courses maximum. | 1 year
  Adverse effects
Objective response comparing lesions' targets according to RECIST criteria, at course n°3 and n°6. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicole TUBIANA-MATHIEU, MD, Principal Investigator — CHU de Limoges, medical oncology department ,02 avenue Martin Luther King 87042 Limoges cedex France
Locations (1):
- CHU Limoges, Limoges, Province, France

REFERENCES:
- [Result] Daher Abdi Z, Lavau-Denes S, Premaud A, Urien S, Sauvage FL, Martin J, Leobon S, Marquet P, Tubiana-Mathieu N, Rousseau A. Pharmacokinetics and exposure-effect relationships of capecitabine in elderly patients with breast or colorectal cancer. Cancer Chemother Pharmacol. 2014 Jun;73(6):1285-93. doi: 10.1007/s00280-014-2466-0. Epub 2014 May 7. PMID 24801171